CLINICAL TRIAL: NCT02792439
Title: America Walks: An Observational Study of Walking Behavior Based on Passive Step Tracking Using a Mobile Phone Application
Brief Title: America Walks: An Observational Study of Walking Behavior Based on Passive Step Tracking
Acronym: AMWALKS
Status: Completed | Type: Observational
Sponsor: TrialX Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 20152782
Record Dates: First submitted 2016-05-27; First posted 2016-06-07 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: Fitness; Health kit; Researchkit; Walking

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
America Walks is an observational research study to determine walking behavior of individuals in the United States. The entire study will be conducted virtually by requiring participants to download a mobile phone application (App), The App will leverage the mobile phone's step count sensor technology to automatically determine participants' daily walking activity. Participation is voluntary. Participants can choose not to participate or choose to participate and then stop participating. Participants decision will not result in any penalty or loss of benefits to which they are entitled.

DETAILED DESCRIPTION:
This will be the first study to measure walking activity using mobile phones. It is well known that physical activity can promote well-being and help prevent several chronic diseases. It is recommended that an individual should do moderate to vigorous walking for 30 minutes or walk approximately 10,000 steps everyday. Several studies have reported measuring walking activity using self-reported surveys, or pedometers in samples ranging from a dozen to a couple of thousand participants. However these studies have largely required participants to enter their walking data manually, either from memory or from pedometer recordings.

With the rapid availability of activity sensors embedded in smart-phones (such as Apple's iPhone version 5S and up and several Google's Android phone models), it is now possible to track physical activity data passively from the end-user and do so for longer durations as individuals have increasingly begun to use their Phones as a continuous device of use.

ELIGIBILITY:
Inclusion Criteria:

* Be at-least 18 years old (self -reported)
* Must reside in the United States (50 states and the District of Columbia); this will be self reported by the participant by entering a zip code which will be checked for valid US zip codes.

Exclusion Criteria:

* Does not have a device that supports Apple HealthKit (iPhone 5s or above) or doesn't not have an Android phone with step count sensors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be residents of the United States with smart phone
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Total step count | 30 days
  This is the total step count from enrollment onwards till user completes 30 days, or quits or till end of study (if the participant continues after 30 days)

SECONDARY OUTCOMES:
Average daily step count (baseline, study) | 30 days
  This will be obtained by averaging the step count data 30 days before enrollment and for the 30 days of the study.
Correlation between perception and actual walking | 4 months
  Calculate the correlation between perceived walking activity as measured by survey items and walking activity as determined by the number of actual steps walked
Total step count (baseline) | 30 days
  The total step count collected from the history on the device (if supported) obtained by the step count data of 30 days before enrollment
Standard Deviation of step count | 4 months
Ranking of cities by daily Average step count | 4 months
  All participants will be grouped by their location and location averages will be ranked

CONTACTS AND LOCATIONS:
Overall Officials: Chintan O Patel, PhD, Principal Investigator — TrialX Inc
Locations (1):
- TrialX Inc, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All study data will be released on http://trialx.com/americawalksstudy in aggregate manner and findings will submitted for publication in academic journals such as the Journal of American Medical Informatics. Any identifiable participant information will not be revealed publicly in any manner whatsoever.

REFERENCES:
- [Background] Tudor-Locke C, Bassett DR Jr. How many steps/day are enough? Preliminary pedometer indices for public health. Sports Med. 2004;34(1):1-8. doi: 10.2165/00007256-200434010-00001. PMID 14715035
- [Background] Bassett DR Jr, Wyatt HR, Thompson H, Peters JC, Hill JO. Pedometer-measured physical activity and health behaviors in U.S. adults. Med Sci Sports Exerc. 2010 Oct;42(10):1819-25. doi: 10.1249/MSS.0b013e3181dc2e54. PMID 20305579
- [Background] Harada ND, Chiu V, King AC, Stewart AL. An evaluation of three self-report physical activity instruments for older adults. Med Sci Sports Exerc. 2001 Jun;33(6):962-70. doi: 10.1097/00005768-200106000-00016. PMID 11404662
- [Background] Bravata DM, Smith-Spangler C, Sundaram V, Gienger AL, Lin N, Lewis R, Stave CD, Olkin I, Sirard JR. Using pedometers to increase physical activity and improve health: a systematic review. JAMA. 2007 Nov 21;298(19):2296-304. doi: 10.1001/jama.298.19.2296. PMID 18029834